CLINICAL TRIAL: NCT01290705
Title: Dosage-dependence of Graded Exercise Therapy in Patients With Patellofemoral Pain Syndrome. A Randomized Controlled Clinical Trial.
Brief Title: Dosage-dependence of Graded Exercise Therapy in Patients With Patellofemoral Pain Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17790
Record Dates: First submitted 2011-02-04; First posted 2011-02-07 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Knee; Anterior Cruciate Ligament; Pain; Patella; Exercise Therapy
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Pain; Patella Fracture

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- high exercise (Experimental): High dose, high repetition exercise therapy, 3 times weekly in 12 weeks
  Interventions: Behavioral: High exercise therapy
- low exercise (Experimental): low dose, low repetition exercise therapy, 3 times weekly in 12 weeks
  Interventions: Behavioral: Low exercise therapy

INTERVENTIONS:
Behavioral: High exercise therapy
  Arms: high exercise
Behavioral: Low exercise therapy
  Arms: low exercise

SUMMARY:
With this study two different therapeutic exercise regimens will be compared in patients with anterior knee pain (patellofemoral pain syndrome, PFPS).

DETAILED DESCRIPTION:
Exercise therapy is widely used in the conservative treatment of patellofemoral pain syndrome (PFPS), but there is still no consensus on recommending any specific rehabilitation program.

This study evaluates two different therapeutic exercise regimens in patients with PFPS and their effect on pain at rest and function.

Supervised exercise therapy will be applied in both groups three times a week over a 3-month period with individually tailored and graded exercise programs, differing between groups in terms of number of exercises, number of repetitions and sets, and time spent on performing aerobic exercises.

ELIGIBILITY:
Inclusion Criteria: Presence of at least 3 symptoms of the following:

Pain when

* Walking stairs
* Squatting
* Running
* Cycling
* Sitting with knees flexed for a prolonged period of time
* Grinding of the patella
* Other positive physical tests (Clarke's test, patellar crepitus, tenderness upon palpation of the posterior surface of the patella, patellar facets or surrounding structures)

Exclusion Criteria:

* Knee osteoarthrosis/ arthritis
* previous knee injury or knee operations
* patellar tendinopathy
* Osgood- Schlatter's disease
* Other defined pathological conditions of the knee

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2007-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Pain measured by a Visual analogue scale (VAS). | Pre-test, post-test (after completed intervention at 3 months) and one year follow-up.
  This scale was illustrated with a 100 mm horizontal line with descriptors "no pain" at the 0 mm mark and "worst pain imaginable" anchoring the 100 mm. Participants were required to place a vertical mark on the horizontal line, representing their average level of pain experienced during the last 24 hours. This was done at rest and provided an illustration of the perceived pain severity, rated in millimetres.

SECONDARY OUTCOMES:
Function measured by a Step-down test and by a modified Functional Index Questionnaire (FIQ). | Pre-test, post-test (at 3 months after completed intervention) and at one year follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Harry Størksen, Study Director — Norwegian University of Science and Technology

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Osteras B, Osteras H, Torstensen TA. Long-term effects of medical exercise therapy in patients with patellofemoral pain syndrome: results from a single-blinded randomized controlled trial with 12 months follow-up. Physiotherapy. 2013 Dec;99(4):311-6. doi: 10.1016/j.physio.2013.04.001. Epub 2013 Jun 10. PMID 23764516
- [Result] Osteras B, Osteras H, Torstensen TA, Vasseljen O. Dose-response effects of medical exercise therapy in patients with patellofemoral pain syndrome: a randomised controlled clinical trial. Physiotherapy. 2013 Jun;99(2):126-31. doi: 10.1016/j.physio.2012.05.009. Epub 2012 Jul 24. PMID 23219636